CLINICAL TRIAL: NCT00767234
Title: Predicting DVT Risk in GI Cancer Patients Using Plasma Biomarkers
Brief Title: Permission to Collect Blood Over Time for Research
Status: Terminated | Type: Observational
Why Stopped: Accrual issues - Low Accrual
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: GI0003; GI0003 (Other: Stanford University); 8502 (Other: Stanford IRB)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer; Gastrointestinal Neoplasms; Colon Rectal Cancer Adenocarcinoma; Esophageal Cancer; Gall Bladder Cancer; Gastric (Stomach) Cancer; Gastrooesophageal Cancer; Gastrointestinal Stromal Tumor (GIST); Hepatobiliary Neoplasm; Liver Carcinoma; Gallbladder Carcinoma; Bile Duct Carcinoma; Carcinoma of the Large Intestine; Anal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Gastrointestinal Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Bile Duct Neoplasms; Colonic Neoplasms; Anus Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Observation — Standard of Care

SUMMARY:
To determine whether biomarkers assessed in blood samples can be used to detect individuals at risk for developing blood clots or worsening of their underlying disease. The ultimate goal of the study is to identify key biomarkers derived from blood that are most characteristic and informative of individuals who will go on to develop a clotting complication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >= 18 years old. There are no ethnic restrictions.
* Active cancers of the GI tract (gastroesophageal, colorectal, or pancreatic-biliary) that have completed TNM staging by the American Joint Committee on Cancer; stage III disease if diagnosed within 2 months and all stage IV disease
* Ability to understand and the willingness to sign a written informed consent document.
* Existing staging CT imaging study

Exclusion Criteria:

* Life expectancy < 6 months
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Known pregnancy or positive urine pregnancy test in pre-menopausal women
* On anticoagulant therapy (heparin, warfarin, direct thrombin inhibitors)
* No CT imaging studies, or contraindications to undergoing CT imaging
* Existing or anticipated need for a tunneled central venous catheter
* Clinic visitation to Stanford Cancer center for secondary consultation purposes only
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active cancers of the GI tract
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Identify Biomarkers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Haruka Itakura, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States